CLINICAL TRIAL: NCT07265570
Title: A Phase IIa, Multicenter, Randomized, Double-blind, Placebo-controlled, Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Efficacy of ISM5411 in Adult Patients With Active Ulcerative Colitis
Brief Title: Study Evaluating ISM5411 Administered Orally to Subjects With Active Ulcerative Colitis (BETHESDA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISM5411-201
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
Keywords: Prolyl hydroxylase (PHD) inhibitor; Ulcerative colitis（UC）; Inflammatory bowel disease (IBD)
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients assigned to Cohort 1 will receive ISM5411 tablets up to 12 weeks. (Experimental)
  Interventions: Drug: ISM5411 tablets
- Patients assigned to Cohort 2 will receive ISM5411 tablets up to 12 weeks. (Experimental)
  Interventions: Drug: ISM5411 tablets
- Patients assigned to Cohort 3 will receive ISM5411 tablets up to 12 weeks. (Experimental)
  Interventions: Drug: ISM5411 tablets
- Patients assigned to Cohort 4 will receive placebo up to 12 weeks. (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISM5411 tablets — Dosage Form: Tablet; Frequency of administration: Orally QD.
  Other Names: Garutadustat
  Arms: Patients assigned to Cohort 1 will receive ISM5411 tablets up to 12 weeks.
Drug: ISM5411 tablets — Dosage Form: Tablet; Frequency of administration: Orally QD.
  Other Names: Garutadustat
  Arms: Patients assigned to Cohort 2 will receive ISM5411 tablets up to 12 weeks.
Drug: ISM5411 tablets — Dosage Form: Tablet ; Frequency of administration: Orally QD.
  Other Names: Garutadustat
  Arms: Patients assigned to Cohort 3 will receive ISM5411 tablets up to 12 weeks.
Drug: Placebo — Dosage Form: Tablet; Frequency of administration: Orally QD.
  Arms: Patients assigned to Cohort 4 will receive placebo up to 12 weeks.

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics and clinical efficacy of ISM5411 in adult patients with active ulcerative colitis.

DETAILED DESCRIPTION:
ISM5411 is a gut-restricted small-molecule prolyl hydroxylase (PHD) inhibitor. It can promote the expression of intestinal mucosal protective genes and maintain the integrity and functions of intestinal barrier together with anti-inflammation. It is expected to become a safe and effective therapy to overcome the shortcomings of traditional simple anti-inflammatory drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who fully understand the content, process and possible adverse events of the study and capable of giving written informed consent form (ICF).
2. Female subjects must be nonpregnancy and nonlactating. Subjects (male or female) are willing to take medically approved effective contraceptive measures from the screening period to 3 months after the last administration and have no sperm or egg donation plan during the study period and within 3 months after the last dose.
3. Male or female between 18 and 75 years of age (inclusive), at the time of signing the ICF.
4. Subject has a diagnosis of UC for at least 3 months prior to screening, and meets the criteria defined in the current protocol.
5. If the subjects have concomitant medication defined in the current protocol, they must meet the relevant criteria to be enrolled.

Exclusion Criteria:

1. Subjects have suspected or diagnosed Crohn's disease (CD), undefined colitis, ischemic colitis, fulminant colitis, toxic megacolon, radiation colitis, gastrointestinal perforation (other than appendicitis or penetrating injury), diverticular disease associated with colitis, enterophthisis, abdominal abscess or fistula, etc.
2. Subjects with previously diagnosed but uneradicated or current gastrointestinal dysplasia.
3. Subjects have received surgery for UC or any other type of major intestinal surgery (i.e., surgical procedure requiring general anesthesia) or are likely to require related surgery during the study.
4. Subjects have evidence of a pathogenic intestinal infection, or have a Clostridium Difficile infection or other intestinal infection within 30 days prior to the screening endoscopy or have tested positive for Clostridium Difficile toxins or other intestinal pathogens at the screening period.
5. Subjects have chronic recurring infection and/or active viral infection that, based on the investigator's clinical assessment, make them an unsuitable candidate for the study.
6. Subjects who are unable to take oral medications and/or have an impact on absorption of medication due to severe malnutrition or disease and surgery, etc., or who are currently receiving or plan to receive total parenteral nutrition (TPN) during the study period.
7. Subjects who have received the relevant treatments defined in the protocol.
8. Subjects with recurrent or disseminated (even if single episode) herpes zoster, or cytomegalovirus infection.
9. Subjects who have the risks of tuberculosis defined in the protocol.
10. Subjects have any of the infection defined in the protocol.
11. Subjects who are known to be allergic to the investigational product or any components of it or who have allergic constitution (allergy to multiple drugs or foods).
12. Subjects have unstable or uncontrolled and clinically significant allergic (except for untreated, asymptomatic, seasonal allergies), hematological, endocrine/metabolic, coagulation, immunologic, pulmonary, cardiovascular, hepatic (expect hepatic steatohepatitis), digestion system (expect UC), genitourinary, psychiatric, oncologic or neurological disease or other medical disorder that would make them ineligible for the study.
13. Subjects have concomitant illness that in the opinion of the investigator, are likely to require systemic glucocorticosteroid therapy during the study (e.g., moderate to severe asthma).
14. Subjects have received major organ surgery (except needle biopsy, tracheotomy, gastrotomy, etc.) or significant trauma within 28 days prior to randomization or is likely to require related surgery during the study.
15. Subjects have history of any malignancy within 5 years of screening, except for successfully treated nonmelanoma skin cancer (NMSC), skin basal cell carcinoma, or localized carcinoma in situ of the cervix.
16. Any abnormal results defined in the protocol were identified during the screening period.
17. Subjects have a clinically significant abnormal ECG at screening, including QTcF > 450 msec for males and > 470 msec for females.
18. Subjects have difficulty in venous blood collection or history of acupuncture syncope reaction or blood phobia.
19. Subjects have contraindications to colonoscopy, including but not limited to gastrointestinal fistulas, early post abdominal surgery, severe coagulopathy, large abdominal aneurysms, or any condition that the investigator determines significantly increases the risk of colonoscopy complications.
20. Subjects have a history of alcohol or drug abuse within 3 months of screening, according to the judgement of the investigator. Alcohol abuse refers to consuming alcohol at least twice per day or more than 14 units of alcohol per week.
21. Subjects are unable to maintain smoking and alcohol abstinence during the study.
22. Subjects have participated in other clinical trials of other drugs or medical devices within 30 days prior to screening period and have already received the investigational product, or are currently participating in another clinical trial of a drug or medical device.
23. Subjects are deemed by the investigator to be inappropriate for the study; or have any condition which would confound or interfere with the evaluation of the safety, tolerability, or PK of the investigational drug; or are unable or unwilling to comply with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
The rate of treatment-emergent adverse events (TEAEs) in each group. | Week1 to Week12.
  To evaluate the safety and tolerability of ISM5411.
The rate of serious adverse events (SAEs) and adverse events (AEs) leading to discontinuation of treatment in each group. | Up to 16 weeks.
  To evaluate the safety and tolerability of ISM5411.
Changes and comparisons of the following data for each group of subjects: vital signs, physical examination, laboratory test(blood routine, blood chemistry, urinalysis, coagulation function, etc.), ECG(Heart rate, RR, PR, QRS,QT, QTcF ), etc. | Up to 16 weeks.
  To evaluate the safety and tolerability of ISM5411.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Week1 to Week12.
  To evaluate pharmacokinetics (PK) of ISM5411 in moderately to severely active UC patients.
Peak plasma time (Tmax) | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.
Area under the plasma concentration-time curve extrapolated from time zero to infinity (AUC0-inf). | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t). | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.
Terminal rate constant (λz) | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.
Elimination half-life (t1/2) | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.
Apparent volume of distribution (Vz/F) | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.
Apparent clearance (CL/F) | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.
Mean residence time (MRT) | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.
Colonic tissue concentration (Ccolon) | Week1 to Week12.
  To evaluate PK of ISM5411 in moderately to severely active UC patients.

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Huizhou First Hospital, Huizhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Second Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - ZhongDa Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Meihekou Central Hospital, Tonghua, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Tai 'an City Central Hospital, Taian, Shandong
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi'an Central Hospital, Xian, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China School of Medicine and West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No